CLINICAL TRIAL: NCT04607746
Title: Prospective Open Label, Pivotal Study of the Accuracy of The CapsoCam Colon (CV-3) in Detecting Colonic Polyps, Using Colonoscopy as the Reference
Brief Title: Pivotal Study of the CapsoCam Colon (CV-3) in Detecting Colonic Polyps, Using Colonoscopy as the Reference
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capso Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CLN-CVI-5794
Record Dates: First submitted 2020-10-23; First posted 2020-10-29 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Colonic Polyp
MeSH Terms: conditions — Colonic Polyps | interventions — Capsule Endoscopes

STUDY DESIGN:
Intervention Model Description: Data collected from this study investigated the first generation CV-3 capsule.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Single arm study (Experimental): Subjects swallows the investigational device and undergoes a colonoscopy
  Interventions: Device: Capsule Endoscope

INTERVENTIONS:
Device: Capsule Endoscope — Capsule endoscope used to view colonic mucosa

SUMMARY:
This study will evaluate the safety and effectiveness of the CapsoCam Colon (CV-3) endoscope system for the detection of colonic polyps.

DETAILED DESCRIPTION:
The first phase of the study investigated the first generation of the capsule. The second generation capsule will be investigated in the final phase of enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. At least 45-75 years of age
2. Committed to undergo a colonoscopy, independent of this study
3. Choose to participate and must have signed the IRB-approved informed consent document and agreed to release colonoscopy images and results report to Sponsor

Exclusion Criteria:

1. Colonoscopy or CT-colonography within the past 5 years that demonstrated no polyps
2. Has contraindication for capsule endoscopy or colonoscopy
3. Subject is suspected or diagnosed with familial adenomatous polyposis, hereditary non polyposis colon cancer, or any high-risk genetic syndrome
4. Subject is suspected or diagnosed with inflammatory bowel disease such as ulcerative colitis or Crohn's disease
5. History of incomplete colonoscopy
6. Type I or uncontrolled II Diabetes (Uncontrolled defined as HbA1C>6.4 within the past 3 months and/or with history of constipation or gastroparesis.)
7. Impaired cardiac function assessed as greater than NYHA Class II
8. History of small- or large-bowel obstructive condition
9. Known history of swallowing disorder, and/or ischemic bowel disease neuropathies and/or radiation enteritis
10. Known history of NSAID enteropathy and stricture resulting from taking NSAIDs on a regular basis that, in the opinion of the Investigator, would put the subject at greater risk for capsule endoscope retention
11. Known allergy to ingredients used in bowel preparation and boosters
12. Daily and/or regular narcotic use
13. Decompensated cirrhosis
14. Prior abdominal radiation therapy
15. Diagnosis of anorexia or bulimia
16. History of or suspicion of any of the following: strictures, volvulus or intestinal obstruction, or internal hernias or abdominal surgeries that the Investigator believes should exclude the patient from study participation
17. Known or suspected megacolon
18. Scheduled to undergo MRI examination within 7 days after ingestion of the capsule
19. Has known slow gastric-emptying time or confirmed diagnosis of gastroparesis
20. Pregnant or nursing or is of child-bearing potential and does not practice medically acceptable methods of contraception. WOCBP must have a negative urine pregnancy test at screening.
21. Unable to follow or tolerate fasting, bowel preparation, and other study procedures
22. Any documented medical or psychological condition or significant concurrent illness which, in the Investigator's opinion, would make it unsafe for the subject to participate in this research study or would affect the validity of the study results
23. Are currently enrolled in an interventional clinical study or currently enrolled in or within the last 30 days, a pharmaceutical clinical study
24. Chronic constipation as defined by <3 bowel movements per week, or the use of routine laxatives (other than fiber) to attain regular bowel movements

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1337 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2025-02-14 (Actual)

PRIMARY OUTCOMES:
Positive Percent Agreement/Negative Percent Agreement | 6 weeks
  1. Positive Percent Agreement (PPA) of study device (SD) with computer assisted detection (CADe) for detecting the presence in a subject of the largest polyp detected by optical colonoscopy (OC) if that polyp is >= 6mm, where a match is considered to have occurred if a polyp detected by the device is assessed as having a size within plus or minus 50% of the size of the polyp detected by OC and as having a location within the same or an adjacent colon segment.
  2. Negative percent agreement (NPA) of the SD with CADe for not detecting any polyp >= 6mm in a subject for whom OC did not detect any polyp >=6mm.

SECONDARY OUTCOMES:
Positive Percent Agreement/Negative Percent Agreement--secondary | 6 weeks
  1. PPA...relying on CADe versus not using CADe for detecting the presence....if that polyp is ≥ 6 mm, where there is a match..
  2. NPA....relying on CADe versus not using CADe for not detecting any polyp ≥ 6 mm in a subject for whom OC did not detect any polyp ≥ 6 mm.
  3. PPA with CADe for detecting the presence...if that polyp is ≥ 10 mm, where there is a match..
  4. NPA with CADe for not detecting any polyp ≥ 10 mm in a subject for whom OC did not detect any polyp ≥ 10 mm.
  5. Sensitivity with CADe for detecting advanced neoplasia & is assessed to be =>10 mm in size.
  6. Specificity with CADe for not detecting any lesion ≥ 10 mm when OC did not detect any advanced neoplasia.
  7. PPA with CADe if that polyp is ≥ 6 mm and < 10 mm
  8. Sensitivity with CADe for polyp ≥ 6 mm.

CONTACTS AND LOCATIONS:
Overall Officials: David Shields, MD, Principal Investigator — Gastroenterology Consultant at San Mateo County Medical Center
Locations (23):
- United States (23):
  - Mayo Clinic, Scottsdale, Arizona
  - Gastro Care Institute, Lancaster, California
  - inSite Digestive Health Care, Los Gatos, California
  - Knowledge Research Center, Orange, California
  - Kaiser Permanente Northern California, San Leandro, California
  - Advanced Research Institute, New Port Richey, Florida
  - Digestive and Liver Center of Florida, Orlando, Florida
  - Advanced Gastroenterology Associates, LLC, Palm Harbor, Florida
  - Advanced Research Institute, St. Petersburg, Florida
  - Digestive Health Services, Downers Grove, Illinois
  - Northshore Center for Gastroenterology, Libertyville, Illinois
  - Suburban Gastroenterology, Naperville, Illinois
  - Southwest Gastroenterology, New Lenox, Illinois
  - Digestive Health Specialists, Chelmsford, Massachusetts
  - West Michigan Clinical Research Center, Wyoming, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Hattiesburg GI Associates, Hattiesburg, Mississippi
  - NY total Medical Care, PC, Brooklyn, New York
  - Gastroenterology Group of Rochester, Rochester, New York
  - Great Lakes Gastroenterology Research, Mentor, Ohio
  - Tri-Cities Gastroenterology, Kingsport, Tennessee
  - Vilo Research Group, Houston, Texas
  - Gastroenterology Consultants of SW Virginia, Roanoke, Virginia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2024-08-01): https://cdn.clinicaltrials.gov/large-docs/46/NCT04607746/Prot_000.pdf